CLINICAL TRIAL: NCT03607539
Title: A Randomized, Double-blinded, Phase III Study of Pemetrexed Plus Platinum Chemotherapy With or Without Sintilimab (IBI308) in First Line Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Subjects (Orient-11)
Brief Title: Efficacy and Safety Evaluation of Sintilimab in Patients With Advanced or Metastatic Non-squamous NSCLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI308C302
Record Dates: First submitted 2018-07-12; First posted 2018-07-31 (Actual); Results first posted 2021-02-16 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — sintilimab; Pemetrexed; Platinum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab in combination with pemetrexed and platinum (Experimental): Injection; dosage form: 10ml: 100mg; frequency: 200mgQ3W (qualer 3 weeks); duration: randomization to the date of the first documented tumor progression per RECIST v1.1 criteria Sintilimab 200mg + pemetrexed/ platinum 4 cycles then Sintilimab 200mg + pemetrexed maintains
  Interventions: Drug: Sintilimab; Drug: Pemetrexed; Drug: Platinum
- Sitilimab Placebo Comparator (Placebo Comparator): placebo 2 vials + pemetrexed/ platinum 4 cycles then Sintilimab 200mg + pemetrexed maintains
  Interventions: Drug: Pemetrexed; Drug: Platinum; Drug: Placebos

INTERVENTIONS:
Drug: Sintilimab — 10 mL:100 mg，200mg，Q3W (qualer 3 weeks), day1, I.V.
  Other Names: IBI308
  Arms: Sintilimab in combination with pemetrexed and platinum
Drug: Pemetrexed — 500mg/m^2; Q3W (qualer 3 weeks), day1, I.V.
Drug: Platinum — Q3W (qualer 3 weeks), day1, I.V.; first 4 cycles.
Drug: Placebos — 10 mL:100 mg，200mg，Q3W (qualer 3 weeks), day1, I.V.
  Arms: Sitilimab Placebo Comparator

SUMMARY:
Efficacy and Safety Evaluation of IBI308 in Patients with advanced or metastatic Non-squamous NSCLC

DETAILED DESCRIPTION:
Sintilimab is expected to increase the PFS from 6 months to 9.2 months. Anti-PD-1 therapy in Chinese non-squamous NSCLC naïve patients will be investigated in this clinical trial.

Additionally the correlation between PD-L1 expression and the response to Sintilimab treatment in Chinese non-squamous NSCLC as well as the role of iRECIST in immune checkpoint inhibitor treatment evaluation will also be assessed.

ELIGIBILITY:
Inclusion criteria

1. Sign written informed consent before any trial-related processes are implemented;
2. Age ≥ 18 years and <75 years;
3. Life expectancy exceeds 3 months;
4. The investigator confirmed at least one measurable lesion according to RECIST 1.1.

   A measurable lesion located in the field of previous radiation therapy or after local treatment may be selected as a target lesion if it is confirmed to have progressed;
5. According to the International Lung Cancer Research Association and the American Association for the Classification of Cancer Classification, the 8th edition of the TNM (Tumor Node Metastasis) staging of lung cancer, a histologically or cytologically confirmed locally advanced (IIIB/IIIC phase) that cannot be treated surgically and cannot undergo radical concurrent chemoradiotherapy, Patients with metastatic or recurrent (stage IV) non-squamous NSCLC;
6. Confirmed for patients with EGFR (Epidermal growth factor receptor) or ALK (Anaplastic lymphoma kinase) targeted therapy (documentary evidence of no tumor EGFR-sensitive mutations and no ALK gene rearrangement)
7. The Eastern Cancer Cooperative Group (ECOG) has a performance score of 0 or 1;
8. Have not received any systematic anti-tumor treatment for advanced disease; The patient may have received adjuvant chemotherapy as long as the disease relapses at least 6 months after the last dose of chemotherapy is completed;
9. Adequate hematologic function, defined as absolute neutrophil count ≥1.5×10^9 /L, platelet count ≥100 ×10^9 /L, hemoglobin ≥9g/dL (no blood transfusion or erythropoietin (EPO) within 7 days) Dependency);
10. Adequate liver function, defined as total bilirubin levels ≤ 1.5 times normal upper limit (ULN) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels ≤ 2.5 times ULN in all patients, or for recorded liver Patients with metastasis, AST and ALT levels ≤ 5 times ULN;
11. Adequate renal function, defined as serum creatinine ≤ 1.5 times ULN or measured or calculated creatinine clearance ≥ 60 ml / min (Cockcroft-Gault formula);
12. Coagulation function is adequate, defined as international normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times normal upper limit (ULN); if the subject is receiving anticoagulant therapy, as long as the PT is used in anticoagulant drugs Within the scope;
13. Female subjects of childbearing age should be negative for urine or serum pregnancy test within 72 hours prior to the first study drug administration (Day 1, Day 1). If the urine pregnancy test results are positive or cannot be confirmed as negative, a blood pregnancy test is required.
14. If there is a risk of conception, male and female patients are required to use high-efficiency contraception (ie, an annual failure rate of less than 1%) and continue until at least 180 days after stopping the trial treatment; Note: If abstinence is the usual lifestyle of the subject and the preferred method of contraception, abstinence can be accepted as a method of contraception.

Exclusion criteria:

1. Histological squamous cell-dominated NSCLC; Mixed cell types must distinguish between dominant cell morphology, and if small cell types are present, the subject is not eligible for inclusion;
2. Currently participating in interventional clinical research or treatment, or receiving other research drugs or using research equipment within 4 weeks before the first dose;
3. Previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or against another stimulatory or synergistic inhibition of T cell receptors [eg CTLA-4 (Cytotoxic T lymphocyte antigen-4), OX-40 (also called CD134, cluster of differentiation134), CD137] agent;
4. Received a traditional Chinese medicine with anti-tumor effect, or an immunomodulatory drug (thymosin, interferon, interleukin) within 2 weeks before the first dose, or received major surgery within 3 weeks before the first dose;
5. Pulmonary radiation therapy of >30 Gy within 6 months prior to the first dose;
6. Completed palliative radiotherapy within 7 days prior to the first dose;
7. Clinical active diverticulitis, abdominal abscess, gastrointestinal obstruction and peritoneal metastasis;
8. Have received a physical organ or blood system transplant;
9. There is clinically uncontrollable pleural effusion/peritoneal effusion;
10. known to have severe allergic reactions (≥3 grade) to the active ingredients of Sintilimab, pemetrexed, cisplatin, carboplatin and or any excipients;
11. Active autoimmune diseases requiring systemic treatment (eg, using a disease-modifying drug, corticosteroid or immunosuppressant) within 2 years prior to the first dose. Alternative therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic treatments;
12. Diagnosis of immunodeficiency or study of systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study.

    Physiological doses of corticosteroids (≤10 mg/day of prednisone or equivalent) are permitted;
13. Has not fully recovered from the toxicity and/or complications caused by any intervention before starting treatment (ie, ≤1 or reaching baseline, excluding fatigue or alopecia);
14. Other malignant tumors were diagnosed within 5 years prior to the first dose, with the exception of radical cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, and/or radically resected carcinoma in situ;
15. Active central nervous system (CNS) metastasis and / or cancerous meningitis. Patients with treated brain metastases who have remained clinically stable for at least 2 weeks and have no new or advanced brain metastases may be enrolled and discontinued hormone therapy 3 days prior to the first study drug. Patients with known untreated, asymptomatic brain metastases can be enrolled, but regular imaging assessments of the brain must be performed.
16. There is a history of (non-infectious) pneumonia requiring steroid therapy or the presence of interstitial lung disease 1 year before the first dose;
17. There are active infections that require systemic treatment;
18. Subjects who are unable or unwilling to receive folic acid or vitamin B12 supplementation;
19. There are known cases of mental illness or substance abuse that may have an impact on compliance with the test requirements;
20. A history of human immunodeficiency virus (HIV) infection (ie, HIV 1/2 antibody positive) is known.
21. Untreated active hepatitis B;

    Note: Controlled (treated) hepatitis B subjects also meet the inclusion criteria if the following criteria are met:

    At least 4 weeks of HBV (Hepatitis B virus) antiviral therapy must have been received prior to the first dose of study drug, and the HBV viral load is <1000 copies/ml (200 IU/ml). Subjects who are receiving HBV therapy and have a viral load of <1000 copies/ml (200 IU/ml) should receive antiviral therapy throughout the study treatment period.

    For subjects with anti-HBc (hepatitis B core antigen)(+), HBsAg(-), anti-HBs(-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but viral reactivation is closely monitored;
22. Active HCV (Hepatitis C virus)-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection);
23. Vaccination of live vaccine within 30 days before the first dose (1st cycle, 1st day); Note: Inactivated virus vaccines for seasonal influenza, injectable drugs are permitted; however, live attenuated influenza vaccines (such as FluMist®) are not allowed for intranasal administration;
24. There may be a history of illness or disease evidence, treatment or laboratory abnormalities that may interfere with the subject's full participation in the study, or the investigator believes that participating in the study is not in the best interests of the subject, including dialysis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — SunYat-senUniversity
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, China

REFERENCES:
- [Derived] Liu T, He J, Wang Y, Yang Y, Zhang L, Shi M, Liu J, Sun D, Wang Z, Fang J, Yu Q, Han B, Cang S, Chen G, Mei X, Yang Z, Huang Y, Fang W, Yang Y, Zhao Y, Zhang L. Health-related quality of life and symptoms in patients with previously untreated, locally advanced or metastatic non-squamous non-small cell lung cancer treated with sintilimab or placebo plus pemetrexed and platinum (ORIENT-11): A randomized, double-blind, phase 3 trial. Lung Cancer. 2025 Feb;200:108108. doi: 10.1016/j.lungcan.2025.108108. Epub 2025 Jan 27. PMID 39884222
- [Derived] Liu Z, Yao Y, Zhao M, Zhao Q, Xue J, Huang Y, Qin S. Radiomics Models Derived From Arterial-Phase-Enhanced CT Reliably Predict Both PD-L1 Expression and Immunotherapy Prognosis in Non-small Cell Lung Cancer: A Retrospective, Multicenter Cohort Study. Acad Radiol. 2025 Jan;32(1):493-505. doi: 10.1016/j.acra.2024.07.028. Epub 2024 Jul 31. PMID 39084935
- [Derived] Zhang L, Wang Z, Fang J, Yu Q, Han B, Cang S, Chen G, Mei X, Yang Z, Stefaniak V, Lin Y, Wang S, Zhang W, Sun L, Yang Y. Final overall survival data of sintilimab plus pemetrexed and platinum as First-Line treatment for locally advanced or metastatic nonsquamous NSCLC in the Phase 3 ORIENT-11 study. Lung Cancer. 2022 Sep;171:56-60. doi: 10.1016/j.lungcan.2022.07.013. Epub 2022 Jul 19. PMID 35917647
- [Derived] Yang Y, Wang Z, Fang J, Yu Q, Han B, Cang S, Chen G, Mei X, Yang Z, Ma R, Bi M, Ren X, Zhou J, Li B, Song Y, Feng J, Li J, He Z, Zhou R, Li W, Lu Y, Wang Y, Wang L, Yang N, Zhang Y, Yu Z, Zhao Y, Xie C, Cheng Y, Zhou H, Wang S, Zhu D, Zhang W, Zhang L. Efficacy and Safety of Sintilimab Plus Pemetrexed and Platinum as First-Line Treatment for Locally Advanced or Metastatic Nonsquamous NSCLC: a Randomized, Double-Blind, Phase 3 Study (Oncology pRogram by InnovENT anti-PD-1-11). J Thorac Oncol. 2020 Oct;15(10):1636-1646. doi: 10.1016/j.jtho.2020.07.014. Epub 2020 Aug 8. PMID 32781263

RESULTS

PARTICIPANT FLOW:
Groups:
- Sintilimab Combination: Sintilimab 200mg, pemetrexed 500mg/m2, cisplatin 75mg/m2 or carboplatin AUC 5 IV infusion q3w for 4 cycles, then sintilimab 200mg, pemetrexed 500mg/m2 IV infusion q3w
- Placebo Combination: Placebo 200mg, pemetrexed 500mg/m2, cisplatin 75mg/m2 or carboplatin AUC 5 IV infusion q3w for 4 cycles, then placebo, pemetrexed 500mg/m2 IV infusion q3w
Period: Overall Study
Arm/Group | Sintilimab Combination | Placebo Combination
Started | 266 | 131
Completed | 0 | 0
Not Completed | 266 | 131

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sintilimab Combination | Placebo Combination | Total
Number analyzed (Participants) | 266 | 131 | 397
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.9 (8.35) | 59.5 (8.73) | 59.8 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 32 | 94
  Male | 204 | 99 | 303
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 266 | 131 | 397
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Programmed Cell Death-Ligand(PD-L1) Tumor Proportion Score(TPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy.
  Participants with a TPS ≥1% were classified as PD-L1 positive and participants with a TPS <1% were classified as PD-L1 negative.
  Participants
    PD-L1 <1% (measured by the tumor proportion score [TPS]) | 85 | 44 | 129
    PD-L1 ≥ 1% (measured by the tumor proportion score[TPS]) | 181 | 87 | 268
Platinum Chemotherapy [Count of Participants; unit: Participants]
  Cisplatin | 71 | 33 | 104
  Carboplatin | 195 | 98 | 293

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Independent Radiographic Review Committee (IRRC)
Description: PFS was defined as the time from randomization to the first documented PD or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD
Time Frame: Trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab Combination | Placebo Combination
Number analyzed (Participants) | 266 | 131
Months | 8.9 [7.1 to 11.3] | 5.0 [4.8 to 6.2]

2. Secondary Outcome: Overall Survival (OS)
Description: The analysis population consisted of all randomized participants.
Time Frame: Trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab Combination | Placebo Combination
Number analyzed (Participants) | 266 | 131
Months | NA [NA to NA] — Median OS and OS range lower and upper limit of 95% CI not reached | NA [11.4 to NA] — Median OS and OS range upper limit of 95% CI not reached

3. Secondary Outcome: Objective Response Rate (ORR) by IRRC Assessment
Description: ORR was defined as the percentage of participants in the analysis population who had a confirmed CR (disappearance of all lesions) or PR (at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1, which was modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The percentage of participants who experienced a confirmed CR or PR according to RECIST 1.1 as assessed by IRC was reported as the ORR
Time Frame: Trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sintilimab Combination | Placebo Combination
Number analyzed (Participants) | 266 | 131
Percentage of Participants | 51.9 [45.70 to 58.02] | 29.8 [22.10 to 38.38]

4. Secondary Outcome: Disease Control Rate (DCR) by IRRC Assessment
Time Frame: Trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Sintilimab Combination | Placebo Combination
Number analyzed (Participants) | 266 | 131
Percentage of Participants | 86.8 [82.18 to 90.66] | 75.6 [67.30 to 82.65]

5. Secondary Outcome: Time to Response (TTR) by IRRC Assessment
Description: TTR was defined as the time of participants from the first treatment administration to the first incidence of a confirmed CR (disappearance of all lesions) or PR (at least a 30% decrease in the sum of diameters [SOD] of target lesions, taking as reference the baseline SOD) according to RECIST 1.1, which was modified for this study to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ. The time from first treatment administration to the first incidence of treatment response was reported as the TTR
Time Frame: Trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Population: The analysis population consisted of all randomized participants.
Measure: Median (Full Range); unit: Months
Arm/Group | Sintilimab Combination | Placebo Combination
Number analyzed (Participants) | 266 | 131
Months | 1.51 [1.2 to 7.0] | 2.63 [1.2 to 5.1]

6. Secondary Outcome: Duration of Response (DOR) by IRRC Assessment
Time Frame: From time of first documented evidence of CR or PR trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sintilimab Combination | Placebo Combination
Number analyzed (Participants) | 266 | 131
Months | NA [7.98 to NA] — Median DOR and DOR range upper limit of 95% CI not reached | 5.52 [4.14 to 10.94]

ADVERSE EVENTS:
Time Frame: Trough Database Cutoff Date of 15-Nov-2019 (Up to approximately 16 months)
Description: The incidence (frequency) and severity (according to NCI CTCAE Version 4.03) of adverse events (AEs). Population: All participants receiving ≥1 dose of randomized study drug. All adverse events, including serious adverse events, will be collected since the consent form is signed until 90th day after last administration of investigation products, either observed by investigator or by the spontaneous reported by subjects.
Arm/Group | Sintilimab Combination | Placebo Combination
All-Cause Mortality (participants affected / at risk) | 51/266 | 39/131
Serious Adverse Events (participants affected / at risk) | 75/266 | 39/131
Other Adverse Events (participants affected / at risk) | 265/266 | 131/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab Combination (N=266) | Placebo Combination (N=131)
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Platelet count decreased (Investigations) | 12 | 8
Lymphocyte count decreased (Investigations) | 3 | 0
Neutrophil count decreased (Investigations) | 3 | 2
White blood cell count decreased (Investigations) | 3 | 2
Acid base balance abnormal (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 12 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 6
Erysipelas (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Purulent pericarditis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Infectious pleural effusion (Infections and infestations) | 0 | 1
Myelitis (Infections and infestations) | 0 | 1
Peripheral nerve infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Pericarditis constrictive (Cardiac disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sintilimab Combination (N=266) | Placebo Combination (N=131)
Neutrophil count decreased (Investigations) | 189 | 82
White blood cell count decreased (Investigations) | 180 | 84
Platelet count decreased (Investigations) | 113 | 41
Aspartate aminotransferase increased (Investigations) | 109 | 51
Alanine aminotransferase increased (Investigations) | 108 | 51
Lymphocyte count decreased (Investigations) | 34 | 10
Gamma-glutamyltransferase increased (Investigations) | 33 | 14
Blood glucose increased (Investigations) | 27 | 8
Weight increased (Investigations) | 24 | 4
Amylase increased (Investigations) | 22 | 13
Blood creatinine increased (Investigations) | 22 | 11
Weight decreased (Investigations) | 22 | 23
Blood alkaline phosphatase increased (Investigations) | 17 | 7
Haemoglobin decreased (Investigations) | 16 | 6
Blood thyroid stimulating hormone increased (Investigations) | 15 | 5
Anaemia (Blood and lymphatic system disorders) | 197 | 103
Nausea (Gastrointestinal disorders) | 108 | 55
Vomiting (Gastrointestinal disorders) | 77 | 41
Constipation (Gastrointestinal disorders) | 71 | 42
Diarrhoea (Gastrointestinal disorders) | 35 | 15
Abdominal distension (Gastrointestinal disorders) | 18 | 12
Decreased appetite (Metabolism and nutrition disorders) | 101 | 41
Hypoalbuminaemia (Metabolism and nutrition disorders) | 53 | 22
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 28 | 16
Hypophagia (Metabolism and nutrition disorders) | 20 | 13
Hypoproteinaemia (Metabolism and nutrition disorders) | 16 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 6
Hypercholesterolaemia (Metabolism and nutrition disorders) | 14 | 10
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 12 | 7
Asthenia (General disorders) | 87 | 42
Pyrexia (General disorders) | 56 | 19
Oedema peripheral (General disorders) | 21 | 9
Chest discomfort (General disorders) | 15 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 16
Productive cough (Respiratory, thoracic and mediastinal disorders) | 19 | 17
Hiccups (Respiratory, thoracic and mediastinal disorders) | 16 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 8
Upper respiratory tract infection (Infections and infestations) | 27 | 12
Pneumonia (Infections and infestations) | 22 | 15
Urinary tract infection (Infections and infestations) | 13 | 8
Rash (Skin and subcutaneous tissue disorders) | 38 | 18
Dizziness (Nervous system disorders) | 28 | 8
Headache (Nervous system disorders) | 15 | 5
Hypoaesthesia (Nervous system disorders) | 12 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 7
Proteinuria (Renal and urinary disorders) | 28 | 13
Haematuria (Renal and urinary disorders) | 12 | 9
Insomnia (Psychiatric disorders) | 30 | 9
Hypothyroidism (Endocrine disorders) | 28 | 14
Hyperthyroidism (Endocrine disorders) | 15 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 20 | 5
Hypertension (Vascular disorders) | 14 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT03607539/Prot_SAP_000.pdf